CLINICAL TRIAL: NCT02784964
Title: A Phase I/II Study to Evaluate the Safety and Efficacy of the Allogeneic Injection of Expanded Adipose-derived Stem Cells to Patients With Knee Osteoarthritis
Brief Title: Adipose-derived Stem Cells (ADSCs) for Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UnicoCell Biomed CO. LTD (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT21
Record Dates: First submitted 2016-05-16; First posted 2016-05-27 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Elixcyte 8mL (Experimental): ADSC 6.4*10^7 cells, allogeneic injection, one time injection on Day 1
  Interventions: Biological: Elixcyte 8 ml
- Hya Joint Plus (Active Comparator): Hya Joint Plus synovial fluid supplement 3mL, SciVision Biotech Inc., one time injection on Day 1
  Interventions: Device: Hya Joint Plus
- Elixcyte 4mL (Experimental): ADSC 3.2*10^7 cells, allogeneic injection, one time injection on Day 1
  Interventions: Biological: Elixcyte 4 ml
- Elixcyte 2mL (Experimental): ADSC 1.6*10^7 cells, allogeneic injection, one time injection on Day 1
  Interventions: Biological: Elixcyte 2 ml

INTERVENTIONS:
Biological: Elixcyte 8 ml — ADSC 6.4*10^7 cells, allogeneic injection
  Arms: Elixcyte 8mL
Device: Hya Joint Plus — Hya Joint Plus synovial fluid supplement 3mL, SciVision Biotech Inc.
  Arms: Hya Joint Plus
Biological: Elixcyte 4 ml — ADSC 3.2*10^7 cells, allogeneic injection
  Arms: Elixcyte 4mL
Biological: Elixcyte 2 ml — ADSC 1.6*10^7 cells, allogeneic injection
  Arms: Elixcyte 2mL

SUMMARY:
1. To assess the safety of allogeneic injection of expanded ADSCs to patients with knee osteoarthritis
2. To assess the efficacy of allogeneic injection of expanded ADSCs to patients with knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-80 years (inclusive)
2. Kellgren-Lawrence grading I-III, as determined by American College of Rheumatology (ACR) criteria for osteoarthritis of the knee
3. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score of 7-17 in the study knee even if treated with chronic doses of non steroidal anti-inflammatory drugs
4. Having provided informed consent

Exclusion Criteria:

1. With previous surgery of articular fracture, ligament reconstruction, meniscal reconstruction, and knee arthroplasty on the target knee joint
2. With previous intra-articular intervention on the target knee joint within past 3 months (e.g. steroid, anaesthetic, sodium hyaluronate)
3. Known or suspected infection of the target knee joint
4. Ascertained hypersensitivity to any component used in the study
5. Administered with systemic anti-inflammatory drugs (e.g. non-steroidal anti-inflammatory drug or steroid ) or topical anti-inflammatory drugs on target knee within 7 days prior to administration in the study
6. With serious prior or ongoing medical conditions (e.g. concomitant illness such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic (e.g. Child-Pugh Class C), psychiatric condition, alcoholism, drug abuse), medical history, physical findings, , or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely affect the safety of the patient
7. With any evidence of malignant disease with life expectancy of less than 1 year
8. Pregnant or lactating women or planning to be pregnant during the study period
9. With body mass index (BMI) greater or equal to 35 kg/m2
10. With joint diseases except knee osteoarthritis considered by investigator not eligible to enter the study
11. With known history of human immunodeficiency virus (HIV) infection.
12. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation
13. With any other serious diseases/medical history considered by the investigator not in the condition to enter the trial
14. Having participated other investigational study within 4 weeks of entering this study
15. With known history of claustrophobia
16. Having any existing active/inactive implanted medical devices, such as cardiac pacemaker, cochlear, intracranial vascular clips or neurostimulator, etc...
17. Having any existing metallic intraocular foreign body

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to post-treatment visit of WOMAC pain score at week 24 after treatment | Weeks 0, 24
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Week 48

SECONDARY OUTCOMES:
Changes from baseline to post-treatment visits of Visual Analogue Scale (VAS) to measure Pain Levels | Weeks 0, 2, 4, 12, 24, 36, 48
Changes from baseline to post-treatment visits of scores of sections in Knee Society Clinical Rating System (KSCRS) Score | Weeks 0, 2, 4, 12, 24, 36, 48
Changes from baseline to post-treatment visits of MRI examination results | Weeks 0, 24, 48, 72, 96
Changes from baseline to post-treatment visits of total score, and sub-scores of all sections in WOMAC | Weeks 0, 2, 4, 12, 36, 48
Total acetaminophen consumption amount during the first 48 weeks and week 48 to week 96 | Week 0, 2, 4, 12, 24, 48, 96
Total non-steroidal anti-inflammatory drug (NSAID) consumption amount during the first 48 weeks and week 48 to week 96 | Weeks 0, 2, 4, 12, 24
Time to subject first time consumes acetaminophen | Weeks 0, 2, 4, 12, 24
Time to subject first time consumes non-steroidal anti-inflammatory drug (NSAID) | Weeks 0, 2, 4, 12, 24
Number of patients with clinically abnormal laboratory values and/or adverse events that are related to treatment | Weeks 0, 2, 4, 12, 24, 36, 48, 72, 96
Number of patients with clinically abnormal vital signs and/or adverse events that are related to treatment | Weeks 0, 2, 4, 12, 24, 36, 48, 72, 96
Changes from baseline to week 96 visit in cartilage thickness in the total femorotibial joint by centralized (independent) imaging interpretation. | Weeks 0, 24, 48, 72, 96

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Han Chang, MD, Principal Investigator — Chang Gung Memorial Hospital; Cheng-Fong Chen, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen CF, Hu CC, Wu CT, Wu HH, Chang CS, Hung YP, Tsai CC, Chang Y. Treatment of knee osteoarthritis with intra-articular injection of allogeneic adipose-derived stem cells (ADSCs) ELIXCYTE(R): a phase I/II, randomized, active-control, single-blind, multiple-center clinical trial. Stem Cell Res Ther. 2021 Oct 30;12(1):562. doi: 10.1186/s13287-021-02631-z. PMID 34717765